CLINICAL TRIAL: NCT01138904
Title: Randomized Phase II Study of FOLFOX Followed by FOLFIRI or Reverse Sequence Treatment in Patients With Advanced or Relapsed Gastric Cancer
Brief Title: FOLFOX Followed by FOLFIRI or Reverse Sequence Treatment in Advanced Gastric Cancer (AGC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A University Hospital (Other)
Collaborators: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sung Yong Oh, Department of internal medicine, Dong-A University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DAUH-AGC-10-1
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; oxaliplatin; irinotecan; sequential treatment
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IROX arm: FOLFIRI -> FOLFOX (Active Comparator): IROX arm: FOLFIRI -> FOLFOX
  FOLFOX REGIMEN
  D1 Oxaliplatin 85mg/m2 + 5DW 500ml MIV over 120min D1,D2 Leucovorin 50mg IV Push D1,D2 5-Fluorouracil 400mg/m2 IV Push D1,D2 5-Fluorouracil 600mg/m2 + 5DW 1000ml MIV over 22hr
  Every 2 weeks
  FOLFILI REGIMEN
  D1 Irinotecan 150mg/m2 + 5DW 500ml MIV over 120min D1,D2 Leucovorin 50mg IV Push D1,D2 5-Fluorouracil 400mg/m2 IV Push D1,D2 5-Fluorouracil 600mg/m2 + 5DW 1000ml MIV over 22hr
  Interventions: Drug: irinotecan, oxaliplatin
- OXIR arm: FOLFIRI -> FOLFOX (Active Comparator): OXIR arm: FOLFIRI -> FOLFOX
  FOLFOX REGIMEN
  D1 Oxaliplatin 85mg/m2 + 5DW 500ml MIV over 120min D1,D2 Leucovorin 50mg IV Push D1,D2 5-Fluorouracil 400mg/m2 IV Push D1,D2 5-Fluorouracil 600mg/m2 + 5DW 1000ml MIV over 22hr
  Every 2 weeks
  FOLFILI REGIMEN
  D1 Irinotecan 150mg/m2 + 5DW 500ml MIV over 120min D1,D2 Leucovorin 50mg IV Push D1,D2 5-Fluorouracil 400mg/m2 IV Push D1,D2 5-Fluorouracil 600mg/m2 + 5DW 1000ml MIV over 22hr
  Interventions: Drug: oxaliplatin, irinotecan

INTERVENTIONS:
Drug: irinotecan, oxaliplatin — OXIR: FOLFOX -> FOLFIRI
  IROX: FOLFIRI -> FOLFOX
  FOLFOX REGIMEN
  D1 Oxaliplatin 85mg/m2 + 5DW 500ml MIV over 120min D1,D2 Leucovorin 50mg IV Push D1,D2 5-Fluorouracil 400mg/m2 IV Push D1,D2 5-Fluorouracil 600mg/m2 + 5DW 1000ml MIV over 22hr
  Every 2 weeks
  FOLFILI REGIMEN
  D1 Irinotecan 150mg/m2 + 5DW 500ml MIV over 120min D1,D2 Leucovorin 50mg IV Push D1,D2 5-Fluorouracil 400mg/m2 IV Push D1,D2 5-Fluorouracil 600mg/m2 + 5DW 1000ml MIV over 22hr
  Every 2 weeks
  Arms: IROX arm: FOLFIRI -> FOLFOX
Drug: oxaliplatin, irinotecan — FOLFOX REGIMEN
  D1 Oxaliplatin 85mg/m2 + 5DW 500ml MIV over 120min D1,D2 Leucovorin 50mg IV Push D1,D2 5-Fluorouracil 400mg/m2 IV Push D1,D2 5-Fluorouracil 600mg/m2 + 5DW 1000ml MIV over 22hr
  Every 2 weeks
  FOLFILI REGIMEN
  D1 Irinotecan 150mg/m2 + 5DW 500ml MIV over 120min D1,D2 Leucovorin 50mg IV Push D1,D2 5-Fluorouracil 400mg/m2 IV Push D1,D2 5-Fluorouracil 600mg/m2 + 5DW 1000ml MIV over 22hr
  Every 2 weeks
  Arms: OXIR arm: FOLFIRI -> FOLFOX

SUMMARY:
FOLFOX* followed by FOLFIRI** or reverse sequence treatment regimen have been used as a standard treatment modality in metastatic colorectal cancer.Oxaliplatin and Irinotecan were used for advanced gastric cancer also. The investigators study was designed to evaluate the safety and efficacy of FOLFOX followed by FOLFIRI or reverse sequence treatment regimen as a first-line and second line therapy for patients with relapsed or metastatic gastric cancer similar with colorectal cancer.

*FOLFOX: oxaliplatin followed by leucovorin before bolus 5-FU followed by continuous infusion 5-FU

**FOLFIRI: irinotecan followed by leucovorin before bolus 5-FU followed by continuous infusion 5-FU

DETAILED DESCRIPTION:
Gastric cancer remains a major public health issue, and is the fourth most common cancer and the second leading cause of cancer deaths worldwide. In Korea, gastric cancer is the most common cancer in men, the second most common cancer in women, and the second leading cause of cancer death. Despite the development of early gastric cancer detection programs, more than two-thirds of patients diagnosed with gastric cancer will develop unresectable disease. Even patients with operable tumors evidence high rates of both local and distant recurrence. In cases of advanced gastric cancer, the median survival rate is 9 to 10 months. Additionally, the overall 5-year survival rate is less than 25% in Korea and Japan.

Several combination regimens of chemotherapy for gastric cancer have been developed, but the survival advantage appears to be marginal, and no worldwide standard regimens have yet been established. Recently, a meta-analysis has been conducted to evaluate the efficacy and tolerability of chemotherapy in patients with advanced gastric cancer. The analysis of chemotherapy versus best supportive care (Hazard Ratio/HR = 0.39, confidence interval (CI) 95% 0.28-0.52) and combination versus single agent, mainly 5-Fluorouracil (5-FU), (HR = 0.83, 95% CI 0.74-0.93) demonstrated significant OS results in favour of chemotherapy and combination chemotherapy. Several chemotherapeutic drugs, including 5-fluorouracil (5-FU), mitomycin C, nitrosoureas, and doxorubicin have evidenced some level of efficacy against advanced gastric cancer. However, the majority of combination chemotherapy regimens for advanced gastric cancer have evidenced overall response rates in a range of 30 to 50% in phase II studies. Furthermore, no new regimens including the use of taxanes or irinotecan have improved either response or survivals in phase II or III trials other than docetaxel, cisplatina and infusional 5-FU (DCF) combination.

Oxaliplatin, a third-generation platinum analogue, is a diaminocyclohexane platinum which forms interstrand DNA adducts, which differ from those formed by cisplatin or carboplatin in terms of their capability to overcome resistance mechanisms. FOLFOX-4 or FOLFOX-6 combination regimen have demonstrated response rate of 38%-50% as a first-line treatment of gastric cancer.

Irinotecan (CPT-11,7-ethyl-10-[4-(1-piperidino)-1-piperidino] is a semi-synthetic plant alkaloid obtained from Camptotheca acuminate of the Nyssaceae family. After conversion to its active metabolite, SN-38, irinotecan acts by inhibiting the eukaryotic enzyme, DNA-topoisomerase I. Single-agent irinotecan has evidenced response rates of 13-23% in cases of advanced gastric cancer. 5-Fluorouracil (5-FU) and Topoisomerase I inhibitor-based regimens have demonstrated a response rate of 20-29%, and have been suggested as a first-line treatment for advanced gastric cancer.

FOLFOX followed by FOLFIRI or reverse sequence treatment regimen have been used as a standard treatment modality in metastatic colorectal cancer.

The study was designed to evaluate the safety and efficacy of FOLFOX followed by FOLFIRI or reverse sequence treatment regimen as a first-line and second line therapy for patients with relapsed or metastatic gastric cancer similar with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric cancer
* No prior chemotherapy for palliative setting
* ECOG PS <3
* Measurable lesion on CT
* adequate kidney function (CCr ≥ 40 ml/min)
* adequate liver function (Transaminase < 3 X upper normal value, Bilirubin < 2 mg%)
* adequate BM function (ANC > 1500/ul, platelet > 75000/ul)
* informed consent

Exclusion Criteria:

* other cancer history
* pregnant or breast feeding
* inadequate general condition for chemotherapy
* allergy to oxaliplatin or irinotecan

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Response rate by RECIST | 6 month after treatment

SECONDARY OUTCOMES:
progression free survival | 1 year after start
overall survival | 2 years after start

CONTACTS AND LOCATIONS:
Overall Officials: HYUK-CHAN KWON, M.D.,Ph.D, Principal Investigator — Dong-A University
Locations (1):
- Sung Yong Oh, Busan, South Korea